CLINICAL TRIAL: NCT02633774
Title: Comparison of Brain Perfusion in Rhythm Control and Rate Control of Persistent Atrial Fibrillation: Prospective Randomized Trial
Brief Title: Comparison of Brain Perfusion in Rhythm Control and Rate Control of Persistent Atrial Fibrillation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2015-0914
Record Dates: First submitted 2015-12-07; First posted 2015-12-17 (Estimated); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Propafenone; apixaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rhythm control group (Active Comparator): 1. Start AAD right after evaluating for LA size, EF, LA thrombus, and presence of CAD during anticoagulation 2. check the echo, brain perfusion CT and K-MOCA on baseline 3. confirm a thrombus through the TEE 4. Cardioversion after 1 month 5. Rhythm FU schedule (2012 ACC/AHA/ESC guidelines) 6. If AF recur, RFCA 7. check the brain perfusion CT, K-MOCA after 3M and 12M
  Interventions: Drug: Propafenone
- Rate control group (Active Comparator): 1. No AAD, just anticoagulation 2. HR control between 60~110bpm (with beta blocker, calcium channel blocker, digoxin) 3. check the echo, brain perfusion CT and K-MOCA on baseline 4. check the brain perfusion CT and K-MOCA after 3M and 12M 5. Without the treatment about antiarrythmia and rhythm control, diffication of rate control, the subject will be drop out for study.
  Interventions: Drug: Apixaban

INTERVENTIONS:
Drug: Propafenone — AAD(antiarrhythmic drug)
  Arms: Rhythm control group
Drug: Apixaban — anti-coagulation
  Arms: Rate control group

SUMMARY:
Atrial fibrillation (AF) is associated with impaired cognitive function (CogF) and/or dementia, but it is unclear whether rhythm control of AF improves CogF or brain perfusion. The hypothesis is rhythm control of AF improves CogF by increasing brain perfusion with hemodynamic amelioration compared to AF state. We will randomize the patients with persistent AF to rhythm control group and rate control group, and check baseline and 3rd month cognitive function (K-MOCA score) and brain perfusion CT. K-MOCA score and brain perfusion CT findings will be compared between rhythm control group and rate control group of persistent AF.

ELIGIBILITY:
Inclusion Criteria:

* Patients with persistent Atrial fibrillation (20~80 years old)
* LA diameter < 55mm
* patients possible to anticoagulation and anti arrhythmic drug

Exclusion Criteria:

* Structural cardiac disease
* Contraindication to brain perfusion CT
* Catheter ablation history for AF, Cardiac surgery
* active internal bleeding
* Impossible to anticoagulation or antiarrhythmic drug
* valvular AF ((MA> GII, Mechanical valve, Mitral valve replacement)
* LVEF < 30%
* With severe medical disease
* Expected survival < 1 year
* Severe alcoholics, drug addiction

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-11; Primary Completion 2020-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
K-MOCA(Korean version of Montreal Cognitive Assessment) | 12 months after the enrollment
Brain perfusion CT | 12 months after the enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Cardiovascular Hospital, Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No